CLINICAL TRIAL: NCT06959420
Title: Knowledge, Attitudes, Perceptions and Behaviors of Healthcare Professionals and the General Population Regarding Vaccination During Febrile Illness
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN322025
Record Dates: First submitted 2025-04-28; First posted 2025-05-06 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Febrile Illness
Keywords: Vaccination; Immunization; Febrile illness; Mild fever; Efficacy; Safety
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthcare professionals: Health professionals who administer vaccines as part of their usual practice.
  Interventions: Other: Questionnaire
- General population: Adults aged 18 years old and over
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Anonymous self-administered questionnaire on the Limesurvey platform.

SUMMARY:
Patients and healthcare professionals often lack adequate information regarding the possibility of vaccinating during febrile illnesses due to limited data. French guidelines on this topic remain vague, placing the responsibility for decision-making on healthcare professionals. This lack of clear guidance, combined with a perceived low urgency for vaccination in such cases, frequently leads to postponements, resulting in missed vaccination opportunities.

By investigating the knowledge, attitudes, perceptions, and behaviors of both patients and healthcare professionals, the investigators can identify obstacles and leverage incentives to promote vaccination during mild febrile illnesses. This approach could help reduce missed opportunities and improve vaccine coverage overall.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare professionals : to administer vaccines as part of their usual practice
* General population: adults aged 18 years old and over.

Exclusion Criteria:

* Healthcare professionals: professionals that do not vaccinate patients in their usual practice.
* General population : individuals under the age of 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People in the general population and healthcare professionals concerned by vaccination.
Sampling Method: Non-Probability Sample
Enrollment: 630 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2025-09-18 (Estimated); Study Completion 2025-09-18 (Estimated)

PRIMARY OUTCOMES:
Population in favour of vaccination during febrile periods | Day 1
  Proportion of the general population and healthcare professionals in favour of vaccination during febrile periods

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Botelho-Nevers, Md PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No